CLINICAL TRIAL: NCT06310083
Title: A Comparative Study of Endoscopic Submucosal Resection Turbinoplasty and Partial Inferior Turbinectomy for Management of Inferior Turbinate Hypertrophy
Brief Title: Endoscopic Submucosal Resection Turbinoplasty VS Turbinectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Nabil Selim (Other)
Responsible Party: Sponsor-Investigator, Ahmed Nabil Selim, Lecturer of otorhinolaryngology, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR for Turbinate Hypertrophy
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Turbinate; Hypertrophy Mucous Membrane
Keywords: turbinoplasty; Turbinectomy; Turbinate Hypertrophy; Endoscopy

STUDY DESIGN:
Intervention Model Description: A total of 40 patients were enrolled in the study. The patients were randomly classified into two groups, with 20 in each group.
  Group A (study group): who applied for Endoscopic submucosal resection Turbinoplasty.
  Group B (control group): Who applied for partial inferior turbinectomy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeons performed the nasal surgery and evaluating postoperative measurable outcomes was blinded about cases who were subjected to Endoscopic submucosal resection Turbinoplasty
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Submucosal Rescetion Turbinoplasty (Active Comparator): participants in this group were applied for Endoscopic submucosal resection Turbinoplasty
  Interventions: Procedure: Submucosal Resection Turbinoplasty Versus Partial Inferior Turbinectomy
- Partial Inferior Turbinectomy (Placebo Comparator): participants in this group were applied for Partial Inferior Turbinectomy
  Interventions: Procedure: Submucosal Resection Turbinoplasty Versus Partial Inferior Turbinectomy

INTERVENTIONS:
Procedure: Submucosal Resection Turbinoplasty Versus Partial Inferior Turbinectomy — The study's Participants Were Randomly classified in two groups Interventional Group, applied for Submucosal Resection Turbinoplasty and the controlled group who were applied for Partial Inferior Turbinectomy

SUMMARY:
The aim of our study is to compare endoscopic submucosal resection Turbinoplasty and partial inferior turbinectomy regarding clinical and radiological evaluation and its possible complications in the treatment of Chronic inferior turbinate hypertrophy.

DETAILED DESCRIPTION:
The inferior turbinate (IT) plays a vital function in nose physiology by regulating the temperature and humidity of inhaled air and filtering foreign particles through the mucociliary clearance system.

One of the most common manifestations of chronic rhinitis is nasal obstruction. Nasal obstruction occurs as a result of submucosal or mucosal hypertrophy associated with increased vascularity of the inferior turbinate.

The location, size, and vasoactive capabilities of the inferior turbinate relegate it as a key player in airway resistance. Multiple pathologic processes may alter the gross and microscopic structure of the inferior turbinates, including septal deviation and inflammatory disorders such as allergic rhinitis, nonallergic rhinitis, and chronic rhinosinusitis. These disorders in turn lead to histological differences in terms of hypertrophy and hyperplasia, distorted cilia, inflammatory cell infiltrates, and mucosal thickening with subsequent macroscopic changes and symptomatic obstruction.

Surgical reduction of the inferior turbinate is warranted to relieve the nasal block caused by the hypertrophied inferior turbinates. Surgical reduction of the inferior turbinate involves removal of the mucosa, soft erectile tissue, and turbinate bone. Different techniques have been applied to increase the nasal airway passage, such as conventional turbinectomy, laser turbinectomy, cryoturbinectomy, electrocautery turbinectomy, conventional Turbinoplasty, microdebrider Turbinoplasty, coblation Turbinoplasty, radiofrequency Turbinoplasty, and ultrasound Turbinoplasty. Conventional turbinectomy (total or partial) is considered very effective in relieving nasal block. Due to the excessive loss of tissue (bone and mucosa), the postoperative complications include excessive bleeding requiring blood transfusion, crusting, pain, and prolonged recovery period. Hence, a more mucosal-friendly approach is preferred; the Turbinoplasty procedure, which resects either soft tissue or bone or both with preservation of the mucosa.

Conventional Turbinoplasty is designed to remove the nonfunctional obstructive part of the turbinate while preserving the functional medial mucosa, which plays the key role in the warming and humidification of air through the nasal passages. Performed endoscopically, inferior Turbinoplasty has the advantage over the other turbinate procedures by preserving sufficient mucosa, while removing adequate obstructed tissue to improve the airway significantly. The other term used for this technique is "submucosal resection", as a reference to its submucosal dissection procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged between 18 and 45 years complaining with a minimum 3-month duration of nasal obstruction combined with clinical findings of inferior turbinate hypertrophy

Exclusion Criteria:

1. Patient's Hemoglobin levels are less than 10gm%.
2. Patients who were Presented with acute upper respiratory tract infection.
3. Patients with other causes of nasal obstruction, e.g.,- allergic nasal polyposis, deviated nasal septum.
4. Patients who have nasal tumors.
5. Patients who had nasal operations before
6. Presence of bleeding disorder.
7. Presence of uncontrolled systemic disease.
8. During the period of menses

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Nasal Obstruction | 3 months
  questionnaire entitled Nasal Obstruction Syndrome Evaluation, known as NOSE score is used to evaluate the improvement in nasal obstruction This score has 5 questions about life quality. Each receives a score from 0 to 4 and these are summed up and multiplied by 20. The total NOSE score ranges from 0 to 100
Nasal Discharge | 3 months
  rhinorrhea conventional visual analogue scale (VAS) is used to evaluate nasal Discharge. Patients were asked to rank their symptoms on a scale of 0-10, with 0 denoting no symptoms and 10 denoting the most severe symptoms, with mild symptoms scoring 0-3, moderate symptoms scoring 4-7, and severe symptoms scoring 8-10
Crustations | 3 months
  an endoscopic score of "Lund and Kennedy" is used to evaluate postoperative Crustations Grade 0 Absence of crustations Grade 1 Mild crustations: partially filling the nasal cavity Grade 2 Severe crustations: fully filling the nasal cavity

SECONDARY OUTCOMES:
intra operative blood loss | intraoperative
  Boezaart surgical field grading scale is used to evaluate intra-operative bleeding (primary), Grade 1 Minimal bleeding, no suction is needed Grade 2 Minimal bleeding, occasional suction is needed Grade 3 Slight bleeding, frequent suction is needed, and surgical field is threatened by bleeding a few seconds after removal of suction Grade 4 Bleeding is moderate, frequent suction is needed, and the surgical field is threatened by bleeding immediately after removal of suction Grade 5 Bleeding is severe, persistent suction is needed, and the surgical field is severely threatened by bleeding that cannot be controlled by suction
Duration of operation (Minutes ) | intraoperative
  Measurement the duration of operation by Minutes
Hyposmia | 3 months
  percentage of patients whose Complaint ( Hyposmia ) Was improved postoperatively

OTHER OUTCOMES:
Size Of Anterior part of Turbinate | Baseline ; 3 months
  Computed Tomography measurements of Anterior part of turbinate pre and postoperatively
Size Of Posterior part of Turbinate | Baseline ; 3 months
  Computed Tomography measurements of posterior part of turbinate pre and postoperatively
Space of Anterior nasal Cavity | Baseline ; 3 months
  Computed Tomography measurements of Anterior part of nasal Cavity pre and postoperatively
Space of posterior nasal Cavity | Baseline ; 3 months
  Computed Tomography measurements of posterior part of nasal Cavity pre and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sabry H Easa, MD, Study Chair — Al-Azhar University Hospital of Assiut
Locations (1):
- Al-Azhar University Hospital of Assiut, Asyut, Egypt

REFERENCES:
- [Background] Al Awad, M. K., & Ali, M. Y. (2022). Inferior Turbinate Hypertrophy Histopathology in Allergic Rhinitis Patients and in Patients with Deviated Nasal Septum. Egyptian Journal of Ear, Nose, Throat and Allied Sciences, 23(23). https://doi.org/10.21608/ejentas.2022.141170.1518
- [Background] Abdullah B, Singh S. Surgical Interventions for Inferior Turbinate Hypertrophy: A Comprehensive Review of Current Techniques and Technologies. Int J Environ Res Public Health. 2021 Mar 26;18(7):3441. doi: 10.3390/ijerph18073441. PMID 33810309
- [Background] Thamboo, A., Ayoub, N., Maul, X., & Nayak, J. (2021a). The Inferior Turbinate: Role in Normal Respiration and Airway Obstruction. In Current Otorhinolaryngology Reports (Vol. 9, Issue 4, 98 pp. 383-388). Springer Science and Business Media B.V. https://doi.org/10.1007/s40136-021- 00370-6
- [Background] Lee KC, Cho JM, Kim SK, Lim KR, Lee SY, Park SS. The Efficacy of Coblator in Turbinoplasty. Arch Craniofac Surg. 2017 Jun;18(2):82-88. doi: 10.7181/acfs.2017.18.2.82. Epub 2017 Jun 26. PMID 28913312
- [Result] Elshipli NA, El-Sisi HE, El-Fattah AMA, Al-Saddeik MAE. Outcome comparison of submucous resection versus combined submucous diathermy and outfracture for treatment of inferior turbinate hypertrophy. Eur Arch Otorhinolaryngol. 2021 Oct;278(10):3827-3837. doi: 10.1007/s00405-021-06663-2. Epub 2021 Feb 13. PMID 33582852
- [Result] Thirugnanamani, R., Sahadevan, S., Ramabhadraiah, A. K., Menon P, A., & M Prabhu, R. (2021). Benefits of Turbinectomy vs Turbinoplasty - A Prospective Study. Bengal Journal of Otolaryngology and Head Neck Surgery, 29(2). https://doi.org/10.47210/bjohns.2021.v29i2.435
- [Result] Amhimmid, R. H., Mohamed, W., Amin, B., Mohamed, A. M., & Odabasha, A. E. (2022). Endoscopic Inferior Turbinoplasty Versus Radiofrequency Ablation for Treatment of Inferior Turbinate Hypertrophy. In The Egyptian Journal of Hospital Medicine (Vol. 88). https://ejhm.journals.ekb.eg/
- [Result] Lund VJ, Kennedy DW. Quantification for staging sinusitis. The Staging and Therapy Group. Ann Otol Rhinol Laryngol Suppl. 1995 Oct;167:17-21. PMID 7574265
- [Derived] Easa SH, Farghaly TM, Elswaby ESS, Selim A. Endoscopic Submucosal Resection Turbinoplasty and Partial Inferior Turbinectomy for Management of Inferior Turbinate Hypertrophy: A Randomized Clinical Trial. Indian J Otolaryngol Head Neck Surg. 2024 Dec;76(6):5080-5090. doi: 10.1007/s12070-024-04926-y. Epub 2024 Aug 8. PMID 39559133